CLINICAL TRIAL: NCT04582500
Title: Low-osmolar Contrast Tagging in Minimal Cathartic CT Colonography
Brief Title: Virtual Colonoscopy Using Omnipaque as a Contrast Agent
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-9791
Record Dates: First submitted 2020-09-30; First posted 2020-10-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer
Keywords: Screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Iohexol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing CTC receiving iohexol: Patients will be recruited from a pool scheduled to undergo screening or diagnostic CTC for clinical purposes. They will be given 50 ml of Iohexol as a oral contrast
  Interventions: Drug: Iohexol

INTERVENTIONS:
Drug: Iohexol — Iohexol (Omnipaque; GE Healthcare, Milwaukee, WI) is a low-osmolar non-ionic iodinated contrast agent that is approved by the FDA for oral use. It is routinely used orally for CT scans of the abdomen and pelvis, and has been used experimentally in CTC. Iohexol is better tolerated by patients and has a better safety profile than hyperosmolar iodinated and barium based contrast agents.
  Other Names: OMNIPAQUE

SUMMARY:
CT colonography (CTC) is a validated screening exam for colorectal cancer. The diagnostic accuracy of CTC depends on the quality of the bowel cleansing and contrast tagging of residual stool and fluid. New bowel preparation media for CTC should be assessed for their efficacy and for patient satisfaction. Iohexol is currently approved by the FDA for oral use for imaging of the gastrointestinal tract. A potential advantage of using iohexol for CTC is that low-and iso-osmolar oral contrast agents have fewer risks than hyperosmolar contrast agents, which make them ideal for use in all patients, especially those who are frail and/or have multiple co-morbidities. For example, hyperosmolar contrast agents that are accidentally aspirated into the lungs during ingestion may result in life-threatening acute pulmonary edema and severe chemical pneumonitis, which is not the case for low- and iso-osmolar contrast agents. It may even be safer to use low- or iso-osmolar contrast agents for patients undergoing CTC on the same day as their incomplete colonoscopy, since they are at risk for aspiration from being sedated for their colonoscopy. Additionally, unlike hyperosmolar contrast agents, low- and iso-osmolar contrast agents do not cause sudden and massive fluid shifts, thus eliminating the risk of dangerous electrolyte imbalances.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer and the second leading cause of cancer-related mortality in the United States when both sexes are combined. Given that the time interval between the appearance of a pre-malignant adenoma and its progression to invasive carcinoma is approximately 5.5 years for polyps >10 mm and 10-15 years for smaller polyps, colorectal cancer is an ideal disease for screening because there is sufficient time to detect and remove pre-malignant adenomas. However, even though screening has been shown to decrease colorectal cancer mortality, only about 60% of people over the age of 50 have had the recommended screening tests.

First introduced in 1994, computed tomography colonography (CTC) is a validated colorectal cancer screening exam by the American Cancer Society. It is a low-radiation dose CT scan of the colon that is performed after bowel preparation and gas insufflation of the colon. CTC has several advantages over optical colonoscopy including less invasiveness, no need for sedation, improved patient comfort, and the ability to identify extracolonic findings. The performance of CTC for polyp detection compares favorably to that of optical colonoscopy and CTC is rapidly gaining acceptance as a screening and diagnostic technique.

For accurate diagnosis in CTC, the colon must be adequately cleansed and any residual stool and fluid must be tagged so that they do not obscure polyps or masses. Patients often find bowel preparation to be the most onerous part of the screening process because it is inconvenient and uncomfortable. Many bowel preparations for CTC and optical colonoscopy require ingestion of large volumes of laxative solutions that can lead to nausea, abdominal pain and diarrhea. Additionally, for CTC, currently the most widely used tagging agents are hyperosmolar iodinated and barium based agents such as diatrizoate meglumine and diatrizoate sodium solution (Gastrografin; Bracco Diagnostics, Monroe Township, NJ), a hyperosmolar ionic iodinated contrast agent. These hyperosmolar agents can also lead to nausea, abdominal pain and diarrhea, and can even result in dangerous electrolyte balances from rapid fluid shifts. Changing the current bowel preparation regimen to improve patient comfort, convenience, and safety would most likely increase patient compliance with CTC.

Iohexol (Omnipaque; GE Healthcare, Milwaukee, WI) is a low-osmolar non-ionic iodinated contrast agent that is approved by the FDA for oral use. It is routinely used orally for CT scans of the abdomen and pelvis, and has been used experimentally in CTC. Iohexol is better tolerated by patients and has a better safety profile than hyperosmolar iodinated and barium based contrast agents.

Study Hypotheses

1. Oral iohexol in conjunction with a minimally cathartic agent results in adequate bowel preparation for CTC.
2. Oral iohexol provides effective tagging of residual stool and fluid in standard screening and diagnostic CTC and same-day CTC following incomplete optical colonoscopy.
3. Oral iohexol is well tolerated by patients in terms of taste, ease of preparation, and side effects.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* able to provide written informed consent

Exclusion Criteria:

* hypersensitivity to iodine-containing compounds,
* pregnant or lactating,
* diuretic therapy, and
* enrollment in other clinical research trials involving investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from a pool scheduled to undergo screening or diagnostic CTC for clinical purposes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
adequate bowel preparation | Within 3 business days of completing CTC
  Two experienced board-certified abdominal imaging radiologists trained in reading CTC will assess percent bowel preparation
Amount of residual fluid and stool | Within 3 business days of completing CTC
  Two experienced board-certified abdominal imaging radiologists trained in reading CTC will assess residual fluid in each of the six segments of the colon (cecum, ascending colon, transverse colon, descending colon, sigmoid colon, and rectum)- Each segment will be scored as - 1 - none, 2 - <25%, 3 - 25-50%, 4: 50-75%, 5: >75%
Efficacy of residual fluid and stool | Within 3 business days of completing CTC
  Two experienced board-certified abdominal imaging radiologists trained in reading CTC will assess residual fluid in each of the six segments of the colon (cecum, ascending colon, transverse colon, descending colon, sigmoid colon, and rectum)- Each segment will be scored as - 1 - none, 2 - <25%, 3 - 25-50%, 4: 50-75%, 5: >75%
Amount of colonic bubbles | Within 3 business days of completing CTC
  Two experienced board-certified abdominal imaging radiologists trained in reading CTC will assess residual fluid in each of the six segments of the colon (cecum, ascending colon, transverse colon, descending colon, sigmoid colon, and rectum)- Each segment will be scored as - 1 - none, 2 - <25%, 3 - 25-50%, 4: 50-75%, 5: >75%
Attenuation of tagged fluid | Within 3 business days of completing CTC
  Two experienced board-certified abdominal imaging radiologists trained in reading CTC will assess residual fluid in each of the six segments of the colon (cecum, ascending colon, transverse colon, descending colon, sigmoid colon, and rectum) It will be recorded in Hounsfield units from Region of Interest (ROI) of fluid in each segment
Patient Satisfaction | immediately after CTC
  Patient satisfaction with Omnipaque 350 as part of their bowel preparation regimen will be assessed with Likert scales in a questionnaire that patient will be asked to fill out after CTC.

SECONDARY OUTCOMES:
Assessing Workflow of incomplete colonoscopies | through study completion, an average of 1 year
  A subset analysis on the workflow of incomplete colonoscopies will also be performed. Specifically those patients who have an incomplete colonoscopy and have a CTC the same day with the Omnipaque regimen and those patients who choose to reattempt or forgo Colorectal cancer screening until a later date.
  The time and resources between those patients who have CTC on the same-day with the Omnipaque regimen after incomplete colonoscopy and the other subset will be compared and determination of the effectiveness of both workflows will be made. This will be used to gauge the productivity for the site.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Yee, MD, FACR, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Background] Muto T, Bussey HJ, Morson BC. The evolution of cancer of the colon and rectum. Cancer. 1975 Dec;36(6):2251-70. doi: 10.1002/cncr.2820360944. PMID 1203876
- [Background] Smith RA, Manassaram-Baptiste D, Brooks D, Doroshenk M, Fedewa S, Saslow D, Brawley OW, Wender R. Cancer screening in the United States, 2015: a review of current American cancer society guidelines and current issues in cancer screening. CA Cancer J Clin. 2015 Jan-Feb;65(1):30-54. doi: 10.3322/caac.21261. Epub 2015 Jan 8. PMID 25581023
- [Background] American Cancer Society. Colorectal Cancer Facts & Figures 2014-2016. Atlanta: American Cancer Society, 2014
- [Background] Thomeer M, Bielen D, Vanbeckevoort D, Dymarkowski S, Gevers A, Rutgeerts P, Hiele M, Van Cutsem E, Marchal G. Patient acceptance for CT colonography: what is the real issue? Eur Radiol. 2002 Jun;12(6):1410-5. doi: 10.1007/s003300101082. Epub 2002 Apr 24. PMID 12042947
- [Background] Levin B, Lieberman DA, McFarland B, Smith RA, Brooks D, Andrews KS, Dash C, Giardiello FM, Glick S, Levin TR, Pickhardt P, Rex DK, Thorson A, Winawer SJ; American Cancer Society Colorectal Cancer Advisory Group; US Multi-Society Task Force; American College of Radiology Colon Cancer Committee. Screening and surveillance for the early detection of colorectal cancer and adenomatous polyps, 2008: a joint guideline from the American Cancer Society, the US Multi-Society Task Force on Colorectal Cancer, and the American College of Radiology. CA Cancer J Clin. 2008 May-Jun;58(3):130-60. doi: 10.3322/CA.2007.0018. Epub 2008 Mar 5. PMID 18322143
- [Background] Lefere PA, Gryspeerdt SS, Dewyspelaere J, Baekelandt M, Van Holsbeeck BG. Dietary fecal tagging as a cleansing method before CT colonography: initial results polyp detection and patient acceptance. Radiology. 2002 Aug;224(2):393-403. doi: 10.1148/radiol.2241011222. PMID 12147834
- [Background] Iannaccone R, Laghi A, Catalano C, Mangiapane F, Lamazza A, Schillaci A, Sinibaldi G, Murakami T, Sammartino P, Hori M, Piacentini F, Nofroni I, Stipa V, Passariello R. Computed tomographic colonography without cathartic preparation for the detection of colorectal polyps. Gastroenterology. 2004 Nov;127(5):1300-11. doi: 10.1053/j.gastro.2004.08.025. PMID 15520999
- [Background] Laghi A, Iannaccone R, Carbone I, Catalano C, Di Giulio E, Schillaci A, Passariello R. Detection of colorectal lesions with virtual computed tomographic colonography. Am J Surg. 2002 Feb;183(2):124-31. doi: 10.1016/s0002-9610(01)00857-1. PMID 11918874
- [Background] Laghi A, Iannaccone R, Carbone I, Catalano C, Panebianco V, Di Giulio E, Schillaci A, Passariello R. Computed tomographic colonography (virtual colonoscopy): blinded prospective comparison with conventional colonoscopy for the detection of colorectal neoplasia. Endoscopy. 2002 Jun;34(6):441-6. doi: 10.1055/s-2002-31999. PMID 12048624
- [Background] Macari M, Bini EJ, Jacobs SL, Lui YW, Laks S, Milano A, Babb J. Significance of missed polyps at CT colonography. AJR Am J Roentgenol. 2004 Jul;183(1):127-34. doi: 10.2214/ajr.183.1.1830127. PMID 15208126
- [Background] Macari M, Bini EJ, Xue X, Milano A, Katz SS, Resnick D, Chandarana H, Krinsky G, Klingenbeck K, Marshall CH, Megibow AJ. Colorectal neoplasms: prospective comparison of thin-section low-dose multi-detector row CT colonography and conventional colonoscopy for detection. Radiology. 2002 Aug;224(2):383-92. doi: 10.1148/radiol.2242011382. PMID 12147833
- [Background] Munikrishnan V, Gillams AR, Lees WR, Vaizey CJ, Boulos PB. Prospective study comparing multislice CT colonography with colonoscopy in the detection of colorectal cancer and polyps. Dis Colon Rectum. 2003 Oct;46(10):1384-90. doi: 10.1007/s10350-004-6755-2. PMID 14530680
- [Background] Pickhardt PJ, Choi JR, Hwang I, Butler JA, Puckett ML, Hildebrandt HA, Wong RK, Nugent PA, Mysliwiec PA, Schindler WR. Computed tomographic virtual colonoscopy to screen for colorectal neoplasia in asymptomatic adults. N Engl J Med. 2003 Dec 4;349(23):2191-200. doi: 10.1056/NEJMoa031618. Epub 2003 Dec 1. PMID 14657426
- [Background] Pickhardt PJ, Taylor AJ, Kim DH, Reichelderfer M, Gopal DV, Pfau PR. Screening for colorectal neoplasia with CT colonography: initial experience from the 1st year of coverage by third-party payers. Radiology. 2006 Nov;241(2):417-25. doi: 10.1148/radiol.2412052007. Epub 2006 Sep 18. PMID 16982816
- [Background] Bayer. Bayer's product. Available via http://www.bayerresources.com.au/resources /uploads/PI/file9348.pdf. Accessed July 15, 2015.
- [Background] U.S. Food and Drug Administration. Omnipaque (iohexol) injection. Available via http:// www.accessdata.fda.gov/drugsatfda_docs/label/2015/018956s095,020608s031lbl.pdf. Accessed July 16, 2015
- [Background] Horton KM, Fishman EK, Gayler B. The use of iohexol as oral contrast for computed tomography of the abdomen and pelvis. J Comput Assist Tomogr. 2008 Mar-Apr;32(2):207-9. doi: 10.1097/RCT.0b013e3180674e44. PMID 18379303
- [Background] McNamara MM, Lockhart ME, Fineberg NS, Berland LL. Oral contrast media for body CT: Comparison of diatrizoate sodium and iohexol for patient acceptance and bowel opacification. AJR Am J Roentgenol. 2010 Nov;195(5):1137-41. doi: 10.2214/AJR.09.3968. PMID 20966319
- [Background] Peterson CM, Lin M, Pilgram T, Heiken JP. Prospective randomized trial of iohexol 350 versus meglumine sodium diatrizoate as an oral contrast agent for abdominopelvic computed tomography. J Comput Assist Tomogr. 2011 Mar-Apr;35(2):202-5. doi: 10.1097/RCT.0b013e3182058e76. PMID 21412090
- [Background] Nagata K, Singh AK, Sangwaiya MJ, Nappi J, Zalis ME, Cai W, Yoshida H. Comparative evaluation of the fecal-tagging quality in CT colonography: barium vs. iodinated oral contrast agent. Acad Radiol. 2009 Nov;16(11):1393-9. doi: 10.1016/j.acra.2009.05.003. Epub 2009 Jul 10. PMID 19596591
- [Background] Kim B, Park SH, Hong GS, Lee JH, Lee JS, Kim HJ, Kim AY, Ha HK. Iohexol versus diatrizoate for fecal/fluid tagging during CT colonography performed with cathartic preparation: comparison of examination quality. Eur Radiol. 2015 Jun;25(6):1561-9. doi: 10.1007/s00330-014-3568-0. Epub 2015 Jan 11. PMID 25576229
- [Background] Hong GS, Park SH, Kim B, Lee JH, Kim JC, Yu CS, Baek S, Lee JS, Kim HJ. Simethicone to prevent colonic bubbles during CT colonography performed with polyethylene glycol lavage and iohexol tagging: a randomized clinical trial. AJR Am J Roentgenol. 2015 Apr;204(4):W429-38. doi: 10.2214/AJR.14.13024. PMID 25794092
- [Background] Zalis ME, Perumpillichira JJ, Magee C, Kohlberg G, Hahn PF. Tagging-based, electronically cleansed CT colonography: evaluation of patient comfort and image readability. Radiology. 2006 Apr;239(1):149-59. doi: 10.1148/radiol.2383041308. PMID 16567485
- [Background] Cai W, Yoshida H, Zalis ME, Nappi JJ, Harris GJ. Informatics in radiology: Electronic cleansing for noncathartic CT colonography: a structure-analysis scheme. Radiographics. 2010 May;30(3):585-602. doi: 10.1148/rg.303095154. Epub 2010 Mar 10. PMID 20219839
- [Background] Fletcher JG, Silva AC, Fidler JL, Cernigliaro JG, Manduca A, Limburg PJ, Wilson LA, Engelby TA, Spencer G, Harmsen WS, Mandrekar J, Johnson CD. Noncathartic CT colonography: Image quality assessment and performance and in a screening cohort. AJR Am J Roentgenol. 2013 Oct;201(4):787-94. doi: 10.2214/AJR.12.9225. PMID 24059367
- [Background] Pollentine A, Ngan-Soo E, McCoubrie P. Acceptability of oral iodinated contrast media: a head-to-head comparison of four media. Br J Radiol. 2013 May;86(1025):20120636. doi: 10.1259/bjr.20120636. PMID 23564884
- [Background] Gryspeerdt S, Lefere P, Herman M, Deman R, Rutgeerts L, Ghillebert G, Baert F, Baekelandt M, Van Holsbeeck B. CT colonography with fecal tagging after incomplete colonoscopy. Eur Radiol. 2005 Jun;15(6):1192-202. doi: 10.1007/s00330-005-2644-x. Epub 2005 Feb 9. PMID 15702335
- [Background] Bielen D, Thomeer M, Vanbeckevoort D, Kiss G, Maes F, Marchal G, Rutgeerts P. Dry preparation for virtual CT colonography with fecal tagging using water-soluble contrast medium: initial results. Eur Radiol. 2003 Mar;13(3):453-8. doi: 10.1007/s00330-002-1755-x. Epub 2002 Nov 14. PMID 12594546
- [Background] Callstrom MR, Johnson CD, Fletcher JG, Reed JE, Ahlquist DA, Harmsen WS, Tait K, Wilson LA, Corcoran KE. CT colonography without cathartic preparation: feasibility study. Radiology. 2001 Jun;219(3):693-8. doi: 10.1148/radiology.219.3.r01jn22693. PMID 11376256
- [Background] Lefere P, Gryspeerdt S, Marrannes J, Baekelandt M, Van Holsbeeck B. CT colonography after fecal tagging with a reduced cathartic cleansing and a reduced volume of barium. AJR Am J Roentgenol. 2005 Jun;184(6):1836-42. doi: 10.2214/ajr.184.6.01841836. PMID 15908539
- [Background] Thomeer M, Carbone I, Bosmans H, Kiss G, Bielen D, Vanbeckevoort D, Van Cutsem E, Rutgeerts P, Marchal G. Stool tagging applied in thin-slice multidetector computed tomography colonography. J Comput Assist Tomogr. 2003 Mar-Apr;27(2):132-9. doi: 10.1097/00004728-200303000-00005. PMID 12703001
- [Background] Zalis ME, Perumpillichira J, Del Frate C, Hahn PF. CT colonography: digital subtraction bowel cleansing with mucosal reconstruction initial observations. Radiology. 2003 Mar;226(3):911-7. doi: 10.1148/radiol.2263012059. Epub 2003 Jan 24. PMID 12601218
- [Background] Iafrate F, Hassan C, Zullo A, Stagnitti A, Ferrari R, Spagnuolo A, Laghi A. CT colonography with reduced bowel preparation after incomplete colonoscopy in the elderly. Eur Radiol. 2008 Jul;18(7):1385-95. doi: 10.1007/s00330-008-0892-2. Epub 2008 Mar 20. PMID 18351357
- [Background] Park SH, Yee J, Kim SH, Kim YH. Fundamental elements for successful performance of CT colonography (virtual colonoscopy). Korean J Radiol. 2007 Jul-Aug;8(4):264-75. doi: 10.3348/kjr.2007.8.4.264. PMID 17673837
- [Background] Johnson B, Hinshaw JL, Robbins JB, Pickhardt PJ. Objective and Subjective Intrapatient Comparison of Iohexol Versus Diatrizoate for Bowel Preparation Quality at CT Colonography. AJR Am J Roentgenol. 2016 Jun;206(6):1202-7. doi: 10.2214/AJR.15.15373. Epub 2016 Mar 24. PMID 27010251